CLINICAL TRIAL: NCT00770835
Title: Effects of Pioglitazone on Endothelial Progenitor Cells in Type 2 Diabetic Patients With Vascular Complications - The SPLENDOR Study.
Brief Title: Efficacy and Safety of Pioglitazone in Treating Subjects With Vascular Complications Associated With Type 2 Diabetes Mellitus.
Acronym: SPLENDOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Medical Director, Takeda Italia Farmaceutici S.p.A.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IT-PIO-109; 2007-003077-44 (EudraCT Number); U1111-1114-3045 (Registry Identifier: WHO)
Record Dates: First submitted 2008-10-08; First posted 2008-10-10 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias | interventions — Pioglitazone; Metformin; Glyburide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone and Metformin QD (Experimental): (along with lifestyle modification)
  Interventions: Drug: Pioglitazone and Metformin
- Glibenclamide and Metformin QD (Active Comparator): (along with lifestyle modification)
  Interventions: Drug: Glibenclamide and Metformin

INTERVENTIONS:
Drug: Pioglitazone and Metformin — Pioglitazone 30 mg, tablets, orally, once daily, metformin stable dose and lifestyle modification for up to 24 weeks.
  Other Names: ACTOS®; AD-4833
  Arms: Pioglitazone and Metformin QD
Drug: Glibenclamide and Metformin — Glibenclamide 10 mg, tablets, orally, once daily and metformin stable dose and lifestyle modification for up to 24 weeks.
  Other Names: Diabeta; Glynase; Micronase; Daonil; Semi-Daonil; Euglucon
  Arms: Glibenclamide and Metformin QD

SUMMARY:
The purpose of this study is to determine the efficacy of pioglitazone compared to glibenclamide, once daily (QD), taken together with metformin and lifestyle modification in type 2 diabetic subjects with cardiovascular disease.

DETAILED DESCRIPTION:
Diabetes is one of the most common chronic diseases worldwide, affecting nearly 200 million people, almost all suffering from Type 2 Diabetes. It is the fourth leading cause of death in developed countries due to the negative impact of the disease on the cardiovascular system. Treatment, aimed to the reduction of this intrinsic cardiovascular risk, is based on tight control of glucose and all coexisting metabolic abnormalities as well as of biomarkers of inflammation and atherogenesis.

Macrovascular complications account for the vast majority of morbidity and mortality in diabetic patients, and there is growing evidence that pathophysiologic mechanisms other than hyperglycemia are responsible. The condition of the vascular endothelium in particular has been shown to effect the health and disease of the cardiovascular system.

The number and function of endothelial progenitor cells correlate inversely with cardiovascular risk factors and may be a surrogate biologic marker for vascular function and cumulative cardiovascular risk.

Pioglitazone is an orally active thiazolidinedione derivative. It is a ligand for peroxisome proliferator-activated receptor-gamma activation that alters transcription of various genes regulating carbohydrate and lipid metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Females must be non-pregnant, non-lactating and post-menopausal.
* A glycosylated hemoglobin level greater than 7.5% and less than 10%.
* Has an age of onset of Type 2 Diabetes greater than 35 years of age.
* Is on metformin monotherapy up to the maximum tolerated daily dose.
* Has a normal or only slightly impaired renal function (a modification of diet in renal disease estimated glomerular filtration rate greater than 60 ml/min/1.73m2.
* Antihypertensives, statins and any other hypolipidemic medications have been initiated at least three months prior to enrollment; no dose modifications are allowed during the study.
* Has one or more cardiovascular comorbidities as follows:

  * stable angina pectoris
  * previous (greater than three months) transient ischemic attack, cerebrovascular accident or carotid atherosclerosis as assessed by bilateral carotid artery ultrasonography
  * peripheral vascular complications documented by a history of claudication or rest pain, ultrasonography or angiography.
* and/or two or more of the following major cardiovascular risk factors:

  * hypertension (blood pressure >130/80 mmHg or treatment)
  * dyslipidemia (low-density lipoprotein-cholesterol >100 mg/dl or treatment and/or high-density lipoprotein-cholesterol <40 mg/dl in men and <45 mg/dl in women or treatment)
  * smoking (>10 cigarettes/day)

Exclusion Criteria:

* Has Type 1 Diabetes.
* Is on insulin therapy.
* Is severely obese defined as a body mass index greater than or equal to 40mg/m2
* Has diabetic retinopathy.
* Has evidence of hepatic dysfunction including liver transaminase greater than three times the upper limit of normal.
* Is unable to remain on a stable dose of the following class of medications 30 days prior to randomization and throughout the six months of the study:

  * antihypertensives
  * statins
  * other hypolipidemic and antiplatelet drugs
* Has a history of alcohol or other drug abuse.
* Has had a new diagnosis of cancer or recurrent cancer within five years of screening.
* Has a need for chronic (greater than two weeks) immunosuppressive therapy.
* Has had heart failure based on the New York Heart Association Functional Class I through IV.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Other antidiabetic drugs (except metformin)
  * Fibrates
  * Rifampicin
  * Glibenclamide interacting drugs, including nonsteroidal anti-inflammatory agents
  * Other drugs that are highly protein bound, including:

    * sulphonamides
    * chloramphenicol
    * probenecid
    * monoamine oxidase inhibitors
    * fluoroquinolones antibiotics
    * oral miconazole
* Has participated in another clinical study within the past three months.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Increase from Baseline in the number of Endothelial Progenitor Cells (CD34+KDR+). | Baseline and Final Visit.

SECONDARY OUTCOMES:
Change from Baseline in Circulating Progenitor Cells Integrated Markers of cardiovascular risk (CD34+). | Baseline and Weeks 12 and 24.
Change from Baseline in Flow Mediated Dilation Integrated Markers of cardiovascular risk. | Baseline and Final Visit.
Modulation of Endothelial Progenitor Cell recruitment (vascular endothelial growth factor, erythropoietin and stromal cell-derived factor-1). | Weeks: 4, 12 and 24.
Measure of Glucose Control (glycosylated hemoglobin and fasting plasma glucose). | Weeks: 4, 12 and 24.
Measure of Lipid Parameters (total lipids, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, triglycerides, apolipoprotein B and apolipoprotein A1). | Weeks: 4, 12 and 24.
Change from Baseline in lipid parameters (free fatty acids and oxidized low-density lipoprotein). | Baseline and Weeks 12 and 24.
Change from Baseline in insulin sensitivity (insulin indexes by 2 hour oral glucose tolerance test with glucose, insulin and C-peptide estimation). | Baseline and Final Visit.
Change from Baseline in Inflammation Markers (high-sensitivity C-reactive protein, IL-6, vascular adhesion molecules (E-selectin, vascular cell adhesion molecule-1), monocyte chemotactic protein-1 and tumor necrosis factor-alpha). | Baseline and Weeks 12 and 24.
Change from Baseline in Adipokines (adiponectin). | Baseline and Weeks 12 and 24.
Change from Baseline in Oxidative Stress (maleic dialdehyde, ferric reducing antioxidant power and lipid hydroperoxide. | Baseline and Weeks 12 and 24.
Urinary albumin excretion. | Weeks: 12 and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (2):
- Italy (2):
  - Padua
  - Pisa

REFERENCES:
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI